CLINICAL TRIAL: NCT07330479
Title: Evaluation of the Efficacy of Ultrasound-Guided Serratus Posterior Superior Intercostal Plane Block For Postoperative Analgesia in Thoracic Surgery
Brief Title: Serratus Posterior Superior Intercostal Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elzem SEN, Assoc. Prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/376
Record Dates: First submitted 2025-12-09; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIPB Group (Experimental): Patients received an ultrasound-guided SPSIPB with 20 mL local anesthetic at the end of surgery.
  Interventions: Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block
- Active Comparator (Active Comparator): Patients received a subcutaneous morphine injection according to institutional standard practice after surgery.
  Interventions: Drug: Subcutaneous Morphine

INTERVENTIONS:
Procedure: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block — Intervention Type: Procedure (Regional Anesthesia) Name: Ultrasound-guided Serratus Posterior Superior Intercostal Plane Block (SPSIPB) Description: A single injection of 20 mL of local anesthetic was administered under ultrasound guidance into the serratus posterior superior intercostal plane at the end of surgery.
  Arms: SPSIPB Group
Drug: Subcutaneous Morphine — Intervention Type: Drug (Morphine) Name: Subcutaneous Morphine Description: Patients received a single subcutaneous injection of morphine (dose according to institutional standard practice) after surgery.
  Arms: Active Comparator

SUMMARY:
Background: Adequate pain control after video-assisted thoracoscopic surgery (VATS) remains a major clinical challenge. Traditional techniques such as thoracic epidural analgesia are effective but limited by potential complications. Interfascial plane blocks have recently gained interest as safer alternatives. The serratus posterior superior intercostal plane block (SPSIPB) is a novel regional anesthesia technique with potential benefits in thoracic surgery.

Objective: The purpose of this study was to evaluate the analgesic efficacy of ultrasound-guided SPSIPB compared with subcutaneous morphine administration in patients undergoing VATS.

Methods: In this prospective, randomized controlled trial, 60 patients scheduled for elective VATS were randomized into two groups: SPSIPB group (n=30) and control group receiving subcutaneous morphine (n=30). The primary outcome was postoperative pain intensity measured by the visual analog scale (VAS) at rest and during coughing. Secondary outcomes included opioid consumption, number of patient-controlled analgesia (PCA) demands, rescue analgesia requirements, and incidence of adverse effects.

DETAILED DESCRIPTION:
Background and Rationale:

Effective postoperative analgesia after thoracic surgery is essential to prevent pulmonary complications, enhance recovery, and improve patient satisfaction. Although thoracic epidural analgesia has traditionally been considered the gold standard, its use is limited due to potential complications such as hypotension, urinary retention, and technical difficulties. With the increased use of minimally invasive thoracic procedures, including video-assisted thoracoscopic surgery (VATS), safer and less invasive analgesic techniques are being explored.

The serratus posterior superior intercostal plane block (SPSIPB) is a newly described regional anesthesia technique that targets the posterior thoracic intercostal nerves. Preliminary evidence suggests that SPSIPB may provide effective postoperative analgesia while minimizing procedure-related risks.

Objective:

The aim of this study was to evaluate the analgesic efficacy and safety of ultrasound-guided SPSIPB compared with subcutaneous morphine injection for postoperative pain management in patients undergoing VATS.

Study Design:

This was a prospective, randomized controlled, single-center clinical trial conducted at Gaziantep University Faculty of Medicine, Department of Anesthesiology. Sixty patients scheduled for elective VATS under general anesthesia were enrolled. After obtaining informed consent, patients were randomly allocated into two groups:

SPSIPB Group (n = 30): Patients received an ultrasound-guided serratus posterior superior intercostal plane block with 20 mL of local anesthetic at the end of surgery.

Control Group (n = 30): Patients received subcutaneous morphine injection according to institutional standard practice.

Outcome Measures:

The primary outcome was postoperative pain intensity assessed by the Visual Analog Scale (VAS) at rest and during coughing at multiple time points within the first 24 hours after surgery. Secondary outcomes included total opioid consumption within 24 hours, the number of patient-controlled analgesia (PCA) demands, the need for rescue analgesia, and the incidence of adverse events such as nausea, vomiting, respiratory depression, or block-related complications.

Significance:

This study will contribute to the growing evidence on interfascial plane blocks in thoracic surgery. If proven effective, SPSIPB may serve as a safe and valuable alternative to conventional analgesic methods, reducing opioid consumption and related side effects in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years
2. American Society of Anesthesiologists (ASA) physical status I-III
3. Scheduled for elective video-assisted thoracoscopic surgery (VATS) under general anesthesia
4. Provision of written informed consent

Exclusion Criteria:

1. Conversion to thoracotomy during surgery
2. Coagulopathy or ongoing anticoagulant therapy
3. Local infection at the injection site
4. Known allergy to local anesthetics or morphine
5. Severe cardiopulmonary disease contraindicating regional anesthesia
6. Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 24 hours after surgery (measured at 0, 2, 4, 8, 16, and 24 hours)
  Pain intensity was assessed using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst pain imaginable) at rest and during coughing.

SECONDARY OUTCOMES:
Total opioid consumption within 24 hours | 24 hours after surgery (cumulative from 0 to 24 hours)
  The cumulative opioid dose administered via patient-controlled analgesia (PCA) and rescue doses was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Şen, Assoc. Prof, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)